CLINICAL TRIAL: NCT04933357
Title: Multimodality- Adapted Dose Modification in Head and Neck Cancer Radiation Therapy Using Functional Imaging
Brief Title: Multimodality- Adapted Dose Modification in Head and Neck Cancer Radiation Therapy ￼
Acronym: MART
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Roa AbdulRahim El-Tagy, assistant lecturer, National Cancer Institute, Egypt
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RO2010-30912
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental)
  Interventions: Radiation: Dose escalation
- Standard dose (Active Comparator)
  Interventions: Radiation: Standard dose

INTERVENTIONS:
Radiation: Dose escalation — Dose escalation to poor responders to achieve dose equivalent more than 80 Gy using SBRT boost
  Arms: Dose escalation
Radiation: Standard dose — Standard dose to good responders to achieve dose equivalent of 70 Gy.
  Arms: Standard dose

SUMMARY:
This is a prospective trial evaluating dose escalation using an SBRT boost to poor- responding tumors by interim functional imaging (PET/CT and fMRI) to improve the local control of HNCSCC.

ELIGIBILITY:
Inclusion Criteria:

* More than or equal to 18 years old. ECOG Performance Scale (0-2). Histological confirmation of SCC of the oral cavity, oropharynx, nasopharynx, hypopharynx or larynx.

Clinical stage II-IVB (AJCC, 8th edition). Multidisciplinary decision of radical radiation or concurrent chemoradiotherapy (CCRT).

Informed consent obtained, signed and dated before specific protocol procedures.

Exclusion Criteria:

* Stage I/II glottic cancer. Patients who underwent surgery for the primary tumor location. Distant metastases. Inability to undergo PET-CT or MRI. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease- free for a minimum of 5 years. Prior radiotherapy to the region of the head and neck that would result in overlap of radiation fields. Any psychological, familial, sociological or geographical condition that hamper compliance with the study and/ or follow up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Loco-regional control of HNSCC patients. | 2 years loco-regional control.

SECONDARY OUTCOMES:
Acute radiation toxicity | During treatment and up to 6 months post treatment.
Comparison between different parameters of PET/CT and fMRI in assessing response to treatment. | 2-4 weeks after start of treatment
Overall survival | 2 years overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Shouman, Study Director — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Cairo, Egypt